CLINICAL TRIAL: NCT04343391
Title: Brief Psychotherapies for Emotional Disorders in Primary and Secondary Care: A Randomized Controlled Trial
Brief Title: Brief Psychotherapies for Emotional Disorders in Primary and Secondary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Jorge Corpas López, Reseracher in Clinical Psychology, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Brief-Psychotherapies
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Emotional Disorder
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Individual Psychotherapy (Experimental): Individual brief psychological intervention by adaptation of the Guide NICE "Common Mental Health Disorders" (ISBN 978-1-84936-585-7) and the unified protocol for the trasndiagnostic treatment of the emotional disorders of Barlow (Boisseau, Farchione, Fairholme, Ellard, y Barlow, 2010). This intervention is provided by clinical psychologist in secondary care.
  Interventions: Behavioral: Brief transdiagnostic cognitive-behavioral therapy
- Brief Group Psychotherapy (Experimental): Group brief psychological intervention by adaptation of the Guide NICE "Common Mental Health Disorders" (ISBN 978-1-84936-585-7) and the unified protocol for the trasndiagnostic treatment of the emotional disorders of Barlow (Boisseau, Farchione, Fairholme, Ellard, y Barlow, 2010). This intervention is provided by clinical psychologist in primary care.
  Interventions: Behavioral: Brief transdiagnostic cognitive-behavioral therapy
- Treatment as usual (Active Comparator): Medication provided by a general practitioner.
  Interventions: Drug: Pharmacological treatment

INTERVENTIONS:
Behavioral: Brief transdiagnostic cognitive-behavioral therapy — Time-limited transdiagnostic evidence-based psychological treatment
  Arms: Brief Group Psychotherapy; Brief Individual Psychotherapy
Drug: Pharmacological treatment — Treatment as usual in PC
  Arms: Treatment as usual

SUMMARY:
The present work aims to develop a randomized clinical trial with a sample of 150 patients diagnosed with at least one of the following emotional disorder: somatoform disorder, panic disorder, generalized anxiety disorder and depression disorder. Participants are tested by several self-reports related to the emocional disorders mentioned in a repeated measures design, pre and post treatment. The investigators think this study will demonstrate that brief psychological treatments should be prioritized over pharmacological treatment for such pathologies in the Primary or Secondary Care context to improve the patient´s quality of life.

DETAILED DESCRIPTION:
Nowadays, the heavy demands placed on health systems exceed the resources in many developed countries. So-called "emotional disorders" and their mostly pharmacological treatment are, in no small part, responsible for this situation. However, research indicates that psychological treatment should be the first step when caring for these types of problems. The investigators expect that the results show that brief psychological therapies are more effective than pharmacological interventions. Moreover, it is expected that brief individual psychotherpay approach delivered in secondary care is more effective than brief group psychotherapy delivered in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Emotional Disorder

Exclusion Criteria:

* Severe mental disorder
* Substance use disorder
* Severe depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-15) | 10 weeks
  The Patient Health Questionnaire-Somatoform Disorder is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-15 is the somatization module, which scores each DSM-IV criteria as "0" (not bothered at all) to "2" (bothered a lot). The more score the more severity.
State-Trait Anxiety Inventory (STAI) | 10 weeks
  The State-Trait Anxiety Inventory is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress AnxietyForm Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level. Internal consistency coefficients for the scale have ranged from .86 to .95; test-retest reliability coefficients have ranged from .65 to .75 over a 2-month interval (Spielberger et al., 1983).
Beck Depression Inventory (BDI-II) | 10 weeks
  The Beck Depression Inventory (second edition) is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults. The BDI-II was revised in 1996 to be more consistent with DSM-IV criteria for depression. For example, individuals are asked to respond to each question based on a two-week time period rather than the one-week timeframe on the BDI. The BDI-II is widely used as an indicator of the severity of depression, but not as a diagnostic tool, and numerous studies provide evidence for its reliability and validity across different populations and cultural groups. The more score the more depression severity.
Patient Health Questionnaire (PHQ-9) | 10 weeks
  The Patient Health Questionnaire-Depression is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The more score the more severity.
Patient Health Questionnaire (PHQ-PD) | 10 weeks
  The Patient Health Questionnaire-Panic Disorder is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-PD is the panic disorder module, which scores each DSM-IV criteria as "yes" or "no". Higher scores mean greater severity of panic disorder.
Generalized Anxiety Disorder score (GAD-7) | 10 weeks
  The Generalized Anxiety Disorder score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD.
Brief Symptom Inventory (BSI-18) | 10 weeks
  The Brief Symptom Inventory contains the three six-item scales somatization, depression, and anxiety as well as the Global Severity Index (GSI), including all 18 items. The BSI-18 is the latest and shortest of the multidimensional versions of the Symptom-Checklist 90-R. The more score the more symptoms patients report.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Córdoba, Córdoba, Córdoba, Spain